CLINICAL TRIAL: NCT07287384
Title: Effects of a Dairy Product Enriched With Lactoferrin on Iron Status of Women With Gestational Diabetes. A Pilot Randomized Controlled Double-blind Trial
Brief Title: Lactoferrin-enriched Dairy Product in Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Simona Bo, Associate Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LACTO_2025
Record Dates: First submitted 2025-10-02; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Gestational Diabetes Mellitus (GDM)
Keywords: Gestational Diabetes Mellitus; Lactoferrin; Iron status in pregnancy
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactoferrin enriched-yogurt (Experimental): In this arm participants were randomized to receved a lactoferrin-enriched yogurt (100mg/125g) twice a day for two months.
  Interventions: Dietary Supplement: Lactoferrin-enriched yogurt supplementation
- Non-enriched yogurt (Other): In this arm participants were randomized to received a non-enriched yogurt(125g) twice a day for two months.
  Interventions: Dietary Supplement: Non-enriched yogurt

INTERVENTIONS:
Dietary Supplement: Lactoferrin-enriched yogurt supplementation — Women were randomized to receive the lactoferrin-enriched yogurt (experimental arm, n=25) - (100mg/125g) 2 times a day for 2 months.Yogurt derived from high-quality cow's milk, with the same color, flavor, and texture as the control group yogurt not enriched with lactoferrin.
  All women of the group received nutritional guidance in accordance with dietary guidelines that accounted for the macronutrient contribution provided by 250g/day of yogurt. The products were provided in unlabeled white plastic cups, distinguishable only by a unique code.
  Arms: Lactoferrin enriched-yogurt
Dietary Supplement: Non-enriched yogurt — Participants were randomized to receved a non-enriched yogurt (125g)- (control arm) twice a day for 2 months. The yogurt was produced from high-quality semi-skimmed cow's milk and It was identical in color, taste, texture, and packaging to the experimental yogurt which conteins lactoferrin. The products were provided in unlabeled white plastic cups, distinguishable only by a unique code.
  Arms: Non-enriched yogurt

SUMMARY:
This pilot double-blind, randomized controlled trial with two parallel arms, was performed to evaluate the change in serum ferritin concentration following consumption of lactoferrin enriched yogurt versus the non-enriched control yogurt in women with GDM.

DETAILED DESCRIPTION:
Lactoferrin is recognized as both effective and safe during pregnancy. Nonetheless, studies specifically investigating its effects in women with GDM are limited.

The primary outcome of this pilot RCT was the change in serum ferritin concentration following the consumption of lactoferrin-enriched yogurt compared with non-enriched control yogurt. Secondary outcomes included changes between the two arms in hemoglobin concentration, hematocrit, red blood cell count, serum iron, transferrin levels, total iron-binding capacity, and transferrin saturation. Additional outcomes were the evaluation of variations in metabolic variables, the occurrence of adverse maternal and neonatal outcomes, and changes in the maternal gut microbiota before and after the intervention

The study began on March 1, 2023, and continued until May 31, 2025. All participants with diagnosis of GDM were recruited according to the inclusion criteria.

Participants received the same dietary counseling and nutritional recommendations aligned with current guidelines by trained registered dieticians. Women were randomized to receive the lactoferrin-enriched yogurt (experimental arm, n=25) and the non-enriched control yogurt (control arm, n=25). Both products were derived from high-quality cow's milk, had the same color, flavor, texture, and were contained in identical unlabeled white 125g plastic cups, each identified solely by a code. The experimental product was enriched with lactoferrin during the manufacturing process (100mg/125g).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GDM confirmed by 75g glucose oral glucose tolerance test (OGTT).
* Caucasian ethnicity, gestational age between 24 and 30 weeks.
* Age >18 and <50 years.
* Body Mass Index (BMI) between 22.5 and 35 kg/m².
* Ability to provide informed consent to participate in the study.

Exclusion Criteria:

* Type 1 diabetes mellitus.
* Allergies to milk proteins or lactose intolerance.
* Known anemia.
* Twin pregnancy.
* Pre-existing iron supplementation exceeding 30 mg/day.
* Insulin therapy at the time of enrollment.
* Any condition or disease requiring specific dietary treatments.
* Concurrent physical or mental conditions requiring pharmacological therapy
* Autoimmune disorders.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change in serum ferritin levels after consumption of lactoferrin-enriched yogurt compared to the non-enriched control yogurt. | 8 weeks - The change in serum ferritin concentration was assessed from baseline to the end of the intervention period.

SECONDARY OUTCOMES:
Changes in Hemoglobin concentration. (HGB) [g/dL] | 8 weeks
  The unit of measure for hemoglobin concentration is grams per deciliter (g/dL).
Occurrence of adverse maternal outcomes [number and percentage of participants] | 8 weeks
  The unit of measure is the number and percentage (%) of participants with at least one adverse maternal event (yes/no).
Changes in Hematocrit values. (HCT) [%] | 8 weeks
  The unit of measure for hematocrit values is percent (%).
Changes in Red Blood Cells count. (RBC) [×10⁶/µL] | 8 WEEKS
  The unit of measure for red blood cell count is ×10⁶ per microliter (µL).
Changes in serum Iron levels. [µg/dL] | 8 weeks
  The unit of measure for serum iron levels is micrograms per deciliter (µg/dL).
Changes in Transferrin levels. [mg/dL] | 8 weeks
  The unit of measure for transferrin levels is milligrams per deciliter (mg/dL).
Change in Total Iron-Binding Capacity (TIBC) [µg/dL] | 8 weeks
  The unit of measure for TIBC is micrograms per deciliter (µg/dL)
Change in Transferrin Saturation. [%] | 8 weeks
  The unit of measure for transferrin saturation is percent (%).
Change in fasting blood glucose concentration (metabolic variables) [mg/dL] | 8 weeks
  The unit of measure for glucose concentration is milligrams per deciliter (mg/dL).
Change in fasting serum insulin levels (metabolic variables) [mIU/L] | 8 weeks
  The unit of measure for insulin is milli-international units per liter (mIU/L).
Occurrence of adverse neonatal outcomes [number and percentage of participants] | At delivery
  The unit of measure is the number and percentage (%) of neonates with at least one adverse neonatal outcome (yes/no).
Changes in the maternal gut microbiota composition. [%] | 8 weeks
  The unit of measure is the relative abundance (%) of bacterial taxa identified by 16S rRNA gene sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Simona Bo, Associate Professor, MD, Principal Investigator — University of Turin, Italy
Locations (1):
- AOU Città della Salute e della Scienza di Torino, University of Torino, Torino., Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT07287384/ICF_000.pdf